CLINICAL TRIAL: NCT04994899
Title: Development of the Aiberry AI Mental Health Screening Platform in a Diverse Population
Brief Title: Aiberry AI Mental Health Screening Platform
Status: Terminated | Type: Observational
Why Stopped: Data collection is no longer necessary
Sponsor: Aiberry, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: Aiberry
Record Dates: First submitted 2021-07-30; First posted 2021-08-06 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-02

CONDITIONS: Depression; Anxiety; Healthy
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aiberry is creating a multi-modal artificial intelligence (AI) platform that analyzes facial, audio and text features to screen for mental illness. This multicenter study will be used to collect data to validate the platform's ability to detect depression and anxiety in a diverse patient population.

DETAILED DESCRIPTION:
Aiberry is developing a proprietary AI platform that leverages machine learning to screen for mental illness using a multi-modal approach that fuses rich visual, audio, text, gestures, and eye gaze information. Our objective in this study is to validate algorithms that predict how individuals will respond to self-report questionnaires used to screen for major depressive disorder (MDD) and general anxiety disorder (GAD). Prior to enrollment, participants will participate in a baseline screening questionnaire to collect demographic information, health history, and current depression severity. If participants meet eligibility requirements and demographic recruitment targets, they will be invited to a single virtual study visit in which they will complete a 10-15 minute recorded interview with a study staff member along with three brief self-report questionnaires: 1) the Quick Inventory of Depression Symptoms Self Report (QIDS-SR-16), 2) the General Anxiety Disorder (GAD-7), and 3) the mini-version of the Mood and Anxiety Questionnaire (mini-MASQ), which will be used as a validity check that participant responses are consistent between this and the previous two questionnaires. We will evaluate how well the AI technology is able to predict self-reported symptoms of depression and anxiety by analyzing facial, audio, and text features from interview videos.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 to 79 years old
* English-speaking

Exclusion Criteria:

* Previous participant in the study, within the last three months
* Individuals unable to verbally respond to standardized questions
* Individuals unable to participate in a virtual visit as they do not have the right hardware (phone/laptop) or no internet connectivity
* Individuals unable to provide consent

Ages: 13 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals with or without prior mental health diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2022-09-22 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Prediction of depression score from a self-report instrument | Single assessment
  Error when predicting depression severity (none, mild, moderate, severe) based on QIDS-SR-16.

SECONDARY OUTCOMES:
Classification of moderate-severe depression | Single assessment
  Accuracy, sensitivity, specificity, and positive and negative predictive value when classifying whether participants meet established cut-off criterion for suspected MDD (QIDS > 10)
Classification of moderate-severe anxiety | Single assessment
  Accuracy, sensitivity, specificity, and positive and negative predictive value when classifying whether participants meet established cut-off criterion for suspected GAD (GAD-7 > 9)
Prediction of anxiety score from a self-report instrument | Single assessment
  Error when predicting anxiety severity (none, mild, moderate, severe) based on GAD-7.

OTHER OUTCOMES:
Prediction of specific anxiety and depression symptoms | Single assessment
  Error when predicting responses to individual items on the QIDS-SR or GAD-7.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Arizona, Tucson, Arizona
  - Georgetown University, Washington D.C., District of Columbia
  - Hapworth Research Inc., New York, New York

IPD SHARING:
Plan to Share IPD: No